CLINICAL TRIAL: NCT03386812
Title: Investigating Bone and Skeletal Muscle Interaction in Men With Prostate Cancer Treated With Androgen Deprivation Therapy.
Brief Title: Investigating Bone and Skeletal Muscle Interaction in Men With Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Charles Y. C. Pak Foundation (Unknown)
Responsible Party: Principal Investigator, Craig D Rubin, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 022017-022
Record Dates: First submitted 2017-12-12; First posted 2017-12-29 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Prostate Cancer
Keywords: androgen deprivation therapy; sarcopenia; bone loss
MeSH Terms: conditions — Prostatic Neoplasms; Sarcopenia; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall goal of this pilot project is to test the hypothesis that a decline in muscle strength precedes the decline in bone strength in men undergoing androgen deprivation therapy (ADT) for prostate cancer. The investigators will measure changes in serum biomarkers involved in muscle-bone crosstalk, anatomic changes in muscle and bone structure and strength that could ultimately contribute to fractures. The findings from this research will inform design of interventions to reduce falls and hip fractures in patients undergoing ADT as well as application to broader populations of at risk patients.

DETAILED DESCRIPTION:
Twenty-five men from urology clinic with prostate cancer will be recruited and enrolled prior to initiating ADT and studied at three time points. Baseline (before first does of ADT), and at approximately weeks 6 and 24 while receiving ADT for prostate cancer. Study measures will be the same during each of three data acquisition time points and include ascertainment of venous blood to determine serum biochemical markers of muscle and bone metabolic activity, MRI and CT imaging studies to assess muscle strength, volume, composition, bone volume, density and strength, and validated tests of muscle strength. Subjects will serve as their own controls.

ELIGIBILITY:
Inclusion Criteria:

• Dx with prostate cancer and planned ADT therapy

Exclusion Criteria:

* Contraindication to MRI
* Limited life expectancy
* Inability to participate in exercise testing
* Severe functional impairment
* Chronic kidney disease 4 or worse
* Hgb < 9
* Use of anti-resorptive agent
* non-English speaking
* Bone metastasis

Ages: 55 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — yes-based on self-representation
Study Population: Men with prostate cancer prior and planning to initiate ADT therapy
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle strength changes with ADT by MRI | 24 weeks
  Absolute muscle fat concentration (% proton density fat fraction) following ADT therapy
Muscle mass changes with ADT treatment | 24 weeks
  Mass of the proximal quadriceps, gluteal and psoas muscles by MRI (cm2)
Myostatin levels following ADT therapy | 24 weeks
  Myostatin ug/ml
Volumetric density following ADT therapy | 24 weeks
  Measure hip bone density in cm3
Gait speed following ADT therapy | 24 weeks
  Gait speed measured in meters per minute
Grip Strength following ADT therapy | 24 weeks
  Grip strength in Kg

CONTACTS AND LOCATIONS:
Overall Officials: Craig Rubin, MD, Principal Investigator — UT Southwestern; Orhan Oz, MD,PhD, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No